CLINICAL TRIAL: NCT05100589
Title: The Effects of PeakATP (Adenosine 5' - Triphosphate Disodium) Supplementation vs. Placebo on Measures of Mood, Reaction Time and Cognitive Performance
Brief Title: Effect of PeakATP on Mood, Reaction Time and Cognition
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Central Florida (Other)
Responsible Party: Principal Investigator, Adam Wells, Associate Professor of Kinesiology, University of Central Florida
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Other
Other Study IDs: STUDY00003272
Record Dates: First submitted 2021-10-07; First posted 2021-10-29 (Actual); Last update posted 2022-08-08 (Actual); Status verified 2022-08

CONDITIONS: Cognitive Change; Mood
Keywords: Adenosine Triphosphate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PeakATP (Experimental): PeakATP formula dissolved in 8 ounces water, taken 30 minutes before breakfast on an empty stomach, or within 30 minutes of waking.
  Interventions: Dietary Supplement: PeakATP
- Placebo (Placebo Comparator): Placebo formula (same as experimental with no PeakATP) dissolved in 8 ounces water, taken 30 minutes before breakfast on an empty stomach, or within 30 minutes of waking.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: PeakATP — Powder - 400mg Peak ATP, maltodextrin, silica-colloidal anhydrous, citric acid anhydrous, sucralose, guar gum
  Arms: PeakATP
Dietary Supplement: Placebo — Powder - maltodextrin, silica-colloidal anhydrous, citric acid anhydrous, sucralose, guar gum
  Arms: Placebo

SUMMARY:
Oral ATP disodium (adenosine 5'- triphosphate disodium) is a commercially available product available alone and as a constituent in a number of sports supplements that is purported to maintain ATP levels and improve performance during high-intensity exercise. Acute deficits in cognitive performance have also been reported in both young adults and children following high-intensity exercise; however, the effects of supplemental ATP on cognitive performance has not been studied.

Goals:

1. To investigate the effect of ATP supplementation versus. placebo on mood, reaction time and cognitive performance before and after an acute bout of fatiguing exercise.
2. To investigate the effect of ATP supplementation versus. placebo on anaerobic performance.

DETAILED DESCRIPTION:
Oral ATP disodium (adenosine 5'- triphosphate disodium) is a commercially available product available alone and as a constituent in a number of sports supplements that is purported to maintain ATP levels during high-intensity exercise. Initial studies providing oral enteric coated ATP disodium displayed no apparent efficacy toward enhancing ATP levels, and subsequent research questioned the bioavailability of enteric coated ATP following oral administration (1,2). However, a recent study demonstrated that ingestion of 400mg uncoated ATP disodium for 15 days prevented decreases in ATP, adenosine diphosphate (ADP), and adenosine monophosphate (AMP) in the bloodstream for up to 30 minutes following high-intensity exercise when compared to placebo (3). Consistent with this, when oral ATP was administered in the form of non-coated ATP disodium, beneficial effects including reduced fatigue (3), improved strength, power, and body composition (5), and enhanced recovery (6) were observed.

Acute deficits in cognitive performance have also been reported in both young adults (6) and children (7) following high-intensity exercise. Cerebral activity is coupled to ATP metabolism, where energy flux is tightly correlated with energy demand (8). Thus, inadequate availability of metabolic resources may lead to acute or long-term cognitive impairments (9) and correspondingly, interventions that sustain ATP levels may have application for attenuating cognitive dysfunction in the face of an acute stressor that challenges brain energy metabolism. Notwithstanding, no study to date has examined the effect of uncoated ATP disodium supplementation on cognitive performance following high-intensity exercise.

Goals:

1. To investigate the the effects of uncoated ATP disodium (PeakATP) on mood (POMS - Profile of mood states questionnaire), psychological stress and cognition (ANAM - Automated Neuropsychological Assessment Metric), reaction time (RT - Dynavision D2 visuomotor tests), and multiple object tracking (MOT - Neurotracker)
2. To examine the effects of uncoated ATP disodium (PeakATP) on end power (mean power during last 30 seconds of 3-minute test), anaerobic working capacity (work above end power), peak power, mean power, time to peak power, fatigue slope (W/sec), rate of fatigue (%), and total work (joules) during a 3-minute all-out cycle ergometer test.

Method:

Randomized, double-blind, placebo controlled cross-over trial comparing the effect of supplementation with Peak ATP versus placebo on mood, reaction time and cognitive performance.

Supplementation will occur over a period of 14 days prior to completion of two separate experimental trials (randomly assigned), with a 14-day washout period in between. An acute dose will also be given during each experimental trial. POMS, RT, MOT and ANAM will be assessed pre- (0) immediately post- (IP) and 60-minutes (60P) post-completion of a 3-minute all-out cycle ergometer test. Anaerobic performance during the 3-minute test will be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Healthy, and ready for physical activity as determined by physical activity readiness questionnaire (PAR-Q+) and medical history questionnaire (MHQ)
* Participants will be required to be recreationally-active (defined according to the American College of Sports Medicine (ACSM) standards of at least 150 minutes exercise per week)
* Participants must currently not be taking and be willing to abstain from creatine or beta-alanine supplementation or be willing to complete a 4-week wash-out period prior to enrolling if taking creatine or beta-alanine and be willing to abstain from supplementing with wither for the duration of the study. This will be verbally confirmed at the beginning of each visit.
* Participant understands the study procedures and signs forms providing informed consent to participate in the study.

Exclusion Criteria:

* Individual does not provide consent to participate in this study.
* Inability to perform physical exercise (determined by MHQ and PAR Q+). That is Answering "Yes" to any question on the PAR-Q +, or having a pre-existing condition such as musculoskeletal injury, back pain, chronic pain etc. that the investigative team perceives will prevent a participant from safely completing the protocol.
* Not currently participating in at least 150 minutes of physical activity per week.
* Currently taking any performance-enhancing drug (determined from health and activity questionnaire)
* Currently taking a nutritional supplement known to improve anerobic performance that requires a wash-out period (e.g., creatine, beta-alanine) and are not willing to undergo a 4-week wash-out period prior to participating.
* Regularly taking any type of prescription or over-the-counter medication, or having any chronic illnesses, which require medical care
* Current known pregnancy

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 35 (Actual)
Dates: Start 2021-10-06 (Actual); Primary Completion 2022-04-19 (Actual); Study Completion 2022-04-19 (Actual)

PRIMARY OUTCOMES:
Mood | Pre (0)
  Assessed via administration of the POMS Questionnaire. 58 words or phrases are presented in a Likert format questionnaire reflecting how the subject feels at the time of completing the questionnaire. Scores range from 0 (Not at all) to 4 (Extremely). Tension, depression, anger, vigor, fatigue, confusion and total mood disturbance (TMD) will be measured.
Mood | Immediately post (IP)
  Assessed via administration of the POMS Questionnaire. 58 words or phrases are presented in a Likert format questionnaire reflecting how the subject feels at the time of completing the questionnaire. Scores range from 0 (Not at all) to 4 (Extremely). Tension, depression, anger, vigor, fatigue, confusion and total mood disturbance (TMD) will be measured.
Mood | 60-minutes post (60P)
  Assessed via administration of the POMS Questionnaire. 58 words or phrases are presented in a Likert format questionnaire reflecting how the subject feels at the time of completing the questionnaire. Scores range from 0 (Not at all) to 4 (Extremely). Tension, depression, anger, vigor, fatigue, confusion and total mood disturbance (TMD) will be measured.
Reaction Time | Pre (0)
  Assessed using the Dynavision D2 visuomotor training device. Subjects are required to recognize and respond as fast as possible to random and sequentially appearing stimuli across the Dynavision apparatus target field.
  Mode A test - The participant will be instructed to successfully identify and strike as many stimuli as possible within 60 seconds with both hands. The number of hits and average reaction time per hit will be assessed.
  Mode B test - The participant will be instructed to successfully identify and strike as many stimuli as possible within 60 seconds with both hands. Additionally, the participant will be required to verbally recite a random 5-digit number that presents on the center screen (t-scope) of the D2. The 5-digit number is presented a total of 11 times throughout the 60-second test, remains for 0.75 seconds and will be randomly generated. The number of hits, misses and the average reaction time per hit will be assessed.
Reaction Time | Immediately post (IP)
  Assessed using the Dynavision D2 visuomotor training device. Subjects are required to recognize and respond as fast as possible to random and sequentially appearing stimuli across the Dynavision apparatus target field.
  Mode A test - The participant will be instructed to successfully identify and strike as many stimuli as possible within 60 seconds with both hands. The number of hits and average reaction time per hit will be assessed.
  Mode B test - The participant will be instructed to successfully identify and strike as many stimuli as possible within 60 seconds with both hands. Additionally, the participant will be required to verbally recite a random 5-digit number that presents on the center screen (t-scope) of the D2. The 5-digit number is presented a total of 11 times throughout the 60-second test, remains for 0.75 seconds and will be randomly generated. The number of hits, misses and the average reaction time per hit will be assessed.
Reaction Time | 60-minutes post (60P)
  Assessed using the Dynavision D2 visuomotor training device. Subjects are required to recognize and respond as fast as possible to random and sequentially appearing stimuli across the Dynavision apparatus target field.
  Mode A test - The participant will be instructed to successfully identify and strike as many stimuli as possible within 60 seconds with both hands. The number of hits and average reaction time per hit will be assessed.
  Mode B test - The participant will be instructed to successfully identify and strike as many stimuli as possible within 60 seconds with both hands. Additionally, the participant will be required to verbally recite a random 5-digit number that presents on the center screen (t-scope) of the D2. The 5-digit number is presented a total of 11 times throughout the 60-second test, remains for 0.75 seconds and will be randomly generated. The number of hits, misses and the average reaction time per hit will be assessed.
Multiple Object Tracking (MOT) | Pre (0)
  Multiple object Tracking (MOT) speed will be assessed via the completion of a CORE assessment using Neurotracker MOT software. The Neurotracker MOT assessment requires participants to track four targets among eight spheres projected within a cube space. The spheres follow a linear trajectory in space, with deviations in trajectory occurring in response to collisions between balls and with the walls of the cube. The CORE assessment includes 20 trials and lasts approx. 6 minutes and challenges attention, visual information processing speed and working memory. The MOT speed threshold, defined as the speed at which the participant correctly identifies all target balls 50% of the time (i.e., the point at which their performance neither improves nor deteriorates) will be determined.
Multiple Object Tracking (MOT) | Immediately post (IP)
  Multiple object Tracking (MOT) speed will be assessed via the completion of a CORE assessment using Neurotracker MOT software. The Neurotracker MOT assessment requires participants to track four targets among eight spheres projected within a cube space. The spheres follow a linear trajectory in space, with deviations in trajectory occurring in response to collisions between balls and with the walls of the cube. The CORE assessment includes 20 trials and lasts approx. 6 minutes and challenges attention, visual information processing speed and working memory. The MOT speed threshold, defined as the speed at which the participant correctly identifies all target balls 50% of the time (i.e., the point at which their performance neither improves nor deteriorates) will be determined.
Multiple Object Tracking (MOT) | 60-minutes post (60P)
  Multiple object Tracking (MOT) speed will be assessed via the completion of a CORE assessment using Neurotracker MOT software. The Neurotracker MOT assessment requires participants to track four targets among eight spheres projected within a cube space. The spheres follow a linear trajectory in space, with deviations in trajectory occurring in response to collisions between balls and with the walls of the cube. The CORE assessment includes 20 trials and lasts approx. 6 minutes and challenges attention, visual information processing speed and working memory. The MOT speed threshold, defined as the speed at which the participant correctly identifies all target balls 50% of the time (i.e., the point at which their performance neither improves nor deteriorates) will be determined.
Symptoms checklist | Pre (0)
  Monitor frequency and severity of subjective symptoms related to a broad spectrum of conditions. The participant is presented with 21 symptoms. The participant is required to rate each symptom (e.g. fatigue, headache, Nausea, numbness/tingling etc. on a scale from 0 (Not Present) to 6 (Severe). Assessed as part of the ANAM.
Symptoms checklist | Immediately post (IP)
  Monitor frequency and severity of subjective symptoms related to a broad spectrum of conditions. The participant is presented with 21 symptoms. The participant is required to rate each symptom (e.g. fatigue, headache, Nausea, numbness/tingling etc. on a scale from 0 (Not Present) to 6 (Severe). Assessed as part of the ANAM.
Sleepiness Scale | 60-minutes post (60P)
  The subject is presented with seven different statements of alertness/sleepiness, ranging from "Feeling very alert, wide awake, and energetic" to "Very sleepy and cannot stay awake much longer." The participant is instructed to select the statement that best matches their current state.
Cognition | Pre (0)
  Response scores from each of seven cognitive assessments administered as part of a battery of tests via Automated Neuropsychological Assessment Metrics (ANAM) computer software. Tests include:
  1. Simple reaction time
  2. Code Substitution
  3. Procedural Reaction Time
  4. Mathematical processing
  5. Matching to sample
  6. Code substitution Delayed
  7. Simple reaction time repeat
Cognition | Immediately post (IP)
  Response scores from each of seven cognitive assessments administered as part of a battery of tests via Automated Neuropsychological Assessment Metrics (ANAM) computer software. Tests include:
  1. Simple reaction time
  2. Code Substitution
  3. Procedural Reaction Time
  4. Mathematical processing
  5. Matching to sample
  6. Code substitution Delayed
  7. Simple reaction time repeat
Cognition | 60-minutes post (60P)
  Response scores from each of seven cognitive assessments administered as part of a battery of tests via Automated Neuropsychological Assessment Metrics (ANAM) computer software. Tests include:
  1. Simple reaction time
  2. Code Substitution
  3. Procedural Reaction Time
  4. Mathematical processing
  5. Matching to sample
  6. Code substitution Delayed
  7. Simple reaction time repeat
Anaerobic performance | During 3-minute test
  Subjects will complete 60 seconds of unloaded cycling at 90 rpm before immediately completing a 3-minute all-out test on a cycle ergometer. Resistance during the test will be set as a function of pedaling rate using a scaling factor based on the power output at a set cadence (70 rpm) being equal to 50% of the difference between the power output at gas exchange threshold (GET) and peak power output assessed during the VO2peak test. End power (mean power during last 30 seconds of 3-minute test), anaerobic working capacity (work above end power), peak power, mean power, time to peak power, fatigue slope (W/sec), rate of fatigue (%), and total work (joules) will be calculated

CONTACTS AND LOCATIONS:
Overall Officials: Adam J Wells, PhD, Principal Investigator — University of Central Florida
Locations (1):
- Kinesiology Research Labs, Orlando, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Du F, Zhu XH, Zhang Y, Friedman M, Zhang N, Ugurbil K, Chen W. Tightly coupled brain activity and cerebral ATP metabolic rate. Proc Natl Acad Sci U S A. 2008 Apr 29;105(17):6409-14. doi: 10.1073/pnas.0710766105. Epub 2008 Apr 28. PMID 18443293
- [Background] Owen L, Sunram-Lea SI. Metabolic agents that enhance ATP can improve cognitive functioning: a review of the evidence for glucose, oxygen, pyruvate, creatine, and L-carnitine. Nutrients. 2011 Aug;3(8):735-55. doi: 10.3390/nu3080735. Epub 2011 Aug 10. PMID 22254121
- [Result] Arts IC, Coolen EJ, Bours MJ, Huyghebaert N, Stuart MA, Bast A, Dagnelie PC. Adenosine 5'-triphosphate (ATP) supplements are not orally bioavailable: a randomized, placebo-controlled cross-over trial in healthy humans. J Int Soc Sports Nutr. 2012 Apr 17;9(1):16. doi: 10.1186/1550-2783-9-16. PMID 22510240
- [Result] Coolen EJ, Arts IC, Bekers O, Vervaet C, Bast A, Dagnelie PC. Oral bioavailability of ATP after prolonged administration. Br J Nutr. 2011 Feb;105(3):357-66. doi: 10.1017/S0007114510003570. Epub 2010 Dec 6. PMID 21129239
- [Result] Purpura M, Rathmacher JA, Sharp MH, Lowery RP, Shields KA, Partl JM, Wilson JM, Jager R. Oral Adenosine-5'-triphosphate (ATP) Administration Increases Postexercise ATP Levels, Muscle Excitability, and Athletic Performance Following a Repeated Sprint Bout. J Am Coll Nutr. 2017 Mar-Apr;36(3):177-183. doi: 10.1080/07315724.2016.1246989. Epub 2017 Jan 12. PMID 28080323
- [Result] Rathmacher JA, Fuller JC Jr, Baier SM, Abumrad NN, Angus HF, Sharp RL. Adenosine-5'-triphosphate (ATP) supplementation improves low peak muscle torque and torque fatigue during repeated high intensity exercise sets. J Int Soc Sports Nutr. 2012 Oct 9;9(1):48. doi: 10.1186/1550-2783-9-48. PMID 23046855
- [Result] Wilson JM, Joy JM, Lowery RP, Roberts MD, Lockwood CM, Manninen AH, Fuller JC, De Souza EO, Baier SM, Wilson SM, Rathmacher JA. Effects of oral adenosine-5'-triphosphate supplementation on athletic performance, skeletal muscle hypertrophy and recovery in resistance-trained men. Nutr Metab (Lond). 2013 Sep 22;10(1):57. doi: 10.1186/1743-7075-10-57. PMID 24330670
- [Result] de Freitas MC, Ricci-Vitor AL, Freire RV, Caperuto EC, Vanderlei LCM, Lira FS, Rossi FE. Oral adenosine 5'-triphosphate supplementation improved hemodynamic and autonomic parameters after exercise in hypertensive women. J Exerc Rehabil. 2018 Aug 24;14(4):671-679. doi: 10.12965/jer.1836256.128. eCollection 2018 Aug. PMID 30276192
- [Result] Sun S, Loprinzi PD, Guan H, Zou L, Kong Z, Hu Y, Shi Q, Nie J. The Effects of High-Intensity Interval Exercise and Hypoxia on Cognition in Sedentary Young Adults. Medicina (Kaunas). 2019 Feb 10;55(2):43. doi: 10.3390/medicina55020043. PMID 30744172
- [Result] Samuel RD, Zavdy O, Levav M, Reuveny R, Katz U, Dubnov-Raz G. The Effects of Maximal Intensity Exercise on Cognitive Performance in Children. J Hum Kinet. 2017 Jun 22;57:85-96. doi: 10.1515/hukin-2017-0050. eCollection 2017 Jun. PMID 28713461